CLINICAL TRIAL: NCT02123004
Title: Comparison of The Influence of Ticagrelor And Clopidogrel on Inflammatory Biomarkers And Vascular Endothelial Function For Patients With ST-Segment Elevation Myocardial Infarction Receiving Emergency Percutaneous Coronary Intervention
Brief Title: Comparison of Ticagrelor And Clopidogrel on Inflammatory Biomarkers And Vascular Endothelial Function
Acronym: TIGERCAVE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jinan Central Hospital (Other)
Responsible Party: Principal Investigator, Su Guohai, Chief Physician, Jinan Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISSBRIL0249; Brilinta-0249 (Other: Study drug trade name and ISS number)
Record Dates: First submitted 2014-04-20; First posted 2014-04-25 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: ST-Segment Elevation Myocardial Infarction
Keywords: ST-Segment Elevation Myocardial Infarction; Percutaneous Coronary Intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor (Experimental): Investigational product/Dosage form and strength/Manufacturer:
  ticagrelor/tablet /90mg/AstraZeneca 180mg loading dose for one day ,then 90mg per day for 4 weeks
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator): Investigational product/Dosage form and strength/Manufacturer:
  clopidogrel/tablet /75mg/Sanofi 300mg loading dose for one day ,then 75mg per day for 4 weeks
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — 180mg loading dose for one day ,and then 90mg per day for 4 weeks
  Other Names: Brilinta
  Arms: Ticagrelor
Drug: Clopidogrel — 300mg loading dose for one day ,and then 75mg per day for 4 weeks
  Other Names: plavix
  Arms: Clopidogrel

SUMMARY:
1. Ticagrelor inhibits inflammation and improves vascular endothelial cell function to a greater extent than clopidogrel in ST-segment elevation myocardial infarction(STEMI) patients receiving percutaneous coronary intervention.
2. Ticagrelor can reduce the serum levels of inflammatory biomarkers both in coronary and in peripheral venous in patients with ST-segment elevation myocardial infarction(STEMI).

DETAILED DESCRIPTION:
Platelet participates in the process of forming and extending atherosclerotic plaques, and it is also a source of inflammatory mediators. This study is a randomized, open-label study, designed to test the hypothesis that ticagrelor inhibits inflammation and improves vascular endothelial cell function to a greater extent than clopidogrel in ST-segment elevation myocardial infarction(STEMI) patients receiving percutaneous coronary intervention. Patients who are scheduled to undergo emergency Percutaneous Coronary Intervention(PCI) will be randomly assigned to receive ticagrelor 180mg for treatment group or clopidogrel 600mg for control group ,then after Percutaneous Coronary Intervention(PCI) treatment group treated with ticagrelor 90mg twice daily while the control group received clopidogrel 75mg once a day . All patients should receive Acetylsalicylic Acid(ASA) 300 mg as a loading dose before Percutaneous Coronary Intervention(PCI) then 100 mg daily unless intolerant. Glycoprotein Ⅱb/Ⅲa receptor antagonists and low-molecular-weight heparin and other additional medication will be directed by the treating cardiologist. All interventions will be performed via the radial approach with the standard technique within 12h after they are involved, and drug-eluting stents will be placed according to stenosis of coronary artery.

The vascular endothelial function will be tested by Circulating Endothelial Cells (CECs) and levels of inflammation will be tested by CD40 ligand (CD40L), C-reactive protein (CRP), and P-selectin to identify that ticagrelor inhibits inflammation and improves vascular endothelial cell function to a greater extent than clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female.
2. Age ≥ 18 years old and <80 years old.
3. Consecutive patients who should be hospitalized with documented evidence of ST-Segment Elevation Myocardial Infarction receiving Percutaneous Coronary Intervention.
4. All patients havepersistent≥0.2 Millivolt ST segment elevation in two or more contiguous precordial leads or ≥0.1 Millivolt ST elevation in two or more contiguous limb leads, with one of the following: persistent chest pain or elevatory of biomarkers of myocardial necrosis.
5. Time from chest pain onset to receiving Percutaneous Coronary Intervention <12 hours.
6. Persistent chest pain <12 hours.
7. Provision of informed consent prior to any study specific procedures.

Exclusion Criteria:

1. Involved in other trials.
2. In recent one year have P 2 Y 12 receptor antagonist drug treatment history or long-term use of immunosuppressive agents.
3. Recurrent myocardial infarction or previous history of Coronary Artery Bypass Graft(CABG) surgery or rescue Percutaneous Coronary Intervention.
4. Active bleeding or bleeding history.
5. With obvious infection and body temperature (axillary temperature) higher than 38.0 ℃.
6. Autoimmune diseases.
7. Malignancies.
8. In recent 6 months have received major surgery.
9. Left ventricular ejection fraction is less than 30%.
10. Life expectancy less than one year.
11. With moderate and severe liver function deterioration.
12. End-stage renal failure.
13. Other conditions that may put the patient at risk or influence study results in the investigators' opinion：eg, increased risk of bradycardiac events; known clinically important thrombocytopenia; known clinically important anemia; severe hemodynamic instability.
14. Other contraindications to investigate products.
15. Any condition that increases the risk for noncompliance or being lost to follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-05 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
CD40 Ligand(CD40l)/C-reactive protein(CRP)/P-selectin and Circulating Endothelial Cells(CECs) | 0 -4 weeks
  The peripheral venous serum level of CD40 Ligand(CD40l)/C-reactive protein(CRP)/P-selectin and Circulating Endothelial Cells(CECs), 0 hour after dosing and 4 weeks after Percutaneous Coronary Intervention(PCI).

SECONDARY OUTCOMES:
CD40 Ligand(CD40l)/C-reactive protein(CRP)/P-selectin and Circulating Endothelial Cells(CECs) | 24hour after dosing
  The peripheral venous serum level of CD40 Ligand(CD40l)/C-reactive protein(CRP)/P-selectin and Circulating Endothelial Cells(CECs), 24hour after dosing and 1 weeks after Percutaneous Coronary Intervention(PCI);
CD40 Ligand(CD40l)/C-reactive protein(CRP)/P-selectin and Circulating Endothelial Cells(CECs) | 1 weeks after Percutaneous Coronary Intervention
  The peripheral venous serum level of CD40 Ligand(CD40l)/C-reactive protein(CRP)/P-selectin and Circulating Endothelial Cells(CECs),24hour after dosing and 1 weeks after Percutaneous Coronary Intervention(PCI);
CD40 Ligand(CD40l)/C-reactive protein(CRP)/P-selectin and Circulating Endothelial Cells(CECs) | 1 hour after dosing
  the coronary serum level of CD40 Ligand(CD40l)/C-reactive protein(CRP)/P-selectin and Circulating Endothelial Cells(CECs),1 hour after dosing;

OTHER OUTCOMES:
Adverse Event | during 4 weeks follow up
  The safety objective of this study in patients will be evaluated by the occurrence of any Adverse Event(AEs) during 4 weeks follow up.Suspected bleeding/reinfarction /rehospitalization /revascularization by Percutaneous Coronary Intervention(PCI) or coronary artery bypass graft (CABG) / sudden death/ stoke /allergic or allergic-like reactions and other adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Su Guohai, Doctor, Principal Investigator — Jinan Central Hospital
Locations (1):
- Jinan Central Hospital, Jinan, Shandong, China

REFERENCES:
- [Derived] Liu P, Wang S, Li K, Yang Y, Man Y, Du F, Wang L, Tian J, Su G. Exosomal microRNA-4516, microRNA-203 and SFRP1 are potential biomarkers of acute myocardial infarction. Mol Med Rep. 2023 Jun;27(6):124. doi: 10.3892/mmr.2023.13010. Epub 2023 May 19. PMID 37203392
- [Derived] Li Z, Li Y, Zhang T, Miao W, Su G. Comparison of the influence of ticagrelor and clopidogrel on inflammatory biomarkers and vascular endothelial function for patients with ST-segment elevation myocardial infarction receiving emergency percutaneous coronary intervention: study protocol for a randomized controlled trial. Trials. 2016 Feb 11;17:75. doi: 10.1186/s13063-016-1168-9. PMID 26865043